CLINICAL TRIAL: NCT04205539
Title: Lymphatic System Health in Alzheimer's Disease
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Pending COVID-19 pandemic
Sponsor: Neurological Associates of West Los Angeles (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20190858
Record Dates: First submitted 2019-12-17; First posted 2019-12-19 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Alzheimer Disease
Keywords: dexmedetomidine; lymphatic system
MeSH Terms: conditions — Alzheimer Disease | interventions — Dexmedetomidine

STUDY DESIGN:
Intervention Model Description: Lumbar punctures will be used to determine Alzheimer's disease status. The subjects will have three fMRI scans: structural T1 and two NOODI DTI scans. The scans take around 45 minutes at no charge to the patients. The dexmedetomidine will be given to the patient after the first DTI scan; this dosage will be congruent with patient height, weight, and medical history. After the subject is asleep, the second DTI scan will be done.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Dexmedetomidine (Experimental): All patients will complete neurocognitive testing inclusive of the Quick Dementia Rating Scale (QDRS) and Repeatable Battery for the Assessment of Neuropsychological Status (RBANS)) to assess cognitive impairment. A Clinical Dementia Rating (CDR) score of 1 or above will be considered dementia. Lumbar punctures will be used to determine Alzheimer's disease status.The subjects will have three fMRI scans: structural T1 and two NOODI DTI scans. The dexmedetomidine will be given to the patient after the first DTI scan with a dosage that will be congruent with patient height, weight, and medical history.
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — This medication will be administered sublingually using an LMA Intranasal Mucosal Atomization Device, which allows the medication to be administered in the form of a spray. Patients will be instructed to keep the medication in their mouth for about 2 minutes, or until fully absorbed. Pulse oximetry and blood pressure will be monitored throughout the duration of treatment. After the subject is asleep, the second DTI scan will be done.
  Other Names: Precedex

SUMMARY:
This study hopes to investigate differences in lymphatic health of patients with Alzheimer's disease by analyzing diffusion-weight images in conscious and sleep states. Dexmedetomidine is a short-acting agent that facilitates a sedated state characterized by slow waves and inhibition of norepinephrine. Conceptually, dexmedetomidine may be preferred to other agents, because it is a short-acting norepinephrine blocker, which could mimic slow wave sleep architecture, opening interstitial spaces, and facilitating plaque removal. Dexmedetomidine may also be preferred given its safety profile among the elderly and acutely ill compared to other anesthetic agents. Sleep will be induced with dexmedetomidine, and interstitial fluid convection will be assessed by measuring free-water diffusion imaging. Freewater diffusion imaging separates out the contributions of extracellular free water and water in the vicinity of cellular tissue; it is used to evaluate abnormalities in extracellular space, such as neuroinflammation, which may contribute to long-term cellular degeneration. This method of analysis could be useful in assessing the lymph systems ability to remove extracellular debris.

DETAILED DESCRIPTION:
The present study is designed as a prospective data analysis of lymphatic system health in Alzheimer's patients and controls. For Phase I trail, 50 patients of any gender with an age range of 18 to 90 who have undergone the outlined procedure will be recruited for inclusion. Patients will be examined by the principle investigator. All patients will complete neurocognitive testing (QDRS and RBANS) to assess cognitive impairment. A CDR score of 1 or above will be considered dementia. Lumbar punctures will be used to determine Alzheimer's disease status. Patients will be offered the option of participating in the study and provided informed consent for neuroimaging. The subjects will have three fMRI scans: structural T1 and two NOODI DTI scans. The scans take around 45 minutes at no charge to the patients. The dexmedetomidine will be given to the patient after the first DTI scan. The dexmedetomidine dosage will be congruent with patient height, weight, and medical history. This medication will be administered sublingually using an LMA Intranasal Mucosal Atomization Device, which allows the medication to be administered in the form of a spray. Patients will be instructed to keep the medication in their mouth for about 2 minutes, or until fully absorbed. Pulse oximetry and blood pressure will be monitored throughout the duration of treatment. After the subject is asleep, the second DTI scan will be done.

ELIGIBILITY:
Inclusion Criteria:

* In order for a subject to be considered for this study, the subject must be willing to comply with the study protocol. They must be between 18 and 90 years old. They must complete neurocognitive testing to assess cognitive impairment (QDRS and RBANS).

Exclusion Criteria:

* Advanced stages of any terminal illness or any active cancer that requires chemotherapy
* Hepatic impairment
* Significant cytopenia
* Cardiovascular, cerebrovascular, and peripheral vascular arterial thrombosis
* Women who are pregnant, may become pregnant, or are breastfeeding
* Any counter indications to dexmedetomidine
* Subjects unable to give informed consent or in vulnerable categories, such as prisoners

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-12-10 (Estimated); Primary Completion 2022-12-10 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
T1 fMRI Imaging | Before dexmedetomidine
  T1-data was collected as a sagittal MPRAGE sequence. T1 images are corrected for field biasing and then skull stripped and linearly registered to standard MNI space. Each patients' T1 image is segmented into 100 cortical and 15 subcortical areas using the Harvard-Oxford Cortical and Subcortical structural atlas. Mean volume is computed for each of these regions for each patient, which can be used for quantitative comparison.
T1 fMRI Imagine | Immediately following administration of dexmedetomidine
  T1-data was collected as a sagittal MPRAGE sequence. T1 images are corrected for field biasing and then skull stripped and linearly registered to standard MNI space. Each patients' T1 image is segmented into 100 cortical and 15 subcortical areas using the Harvard-Oxford Cortical and Subcortical structural atlas. Mean volume is computed for each of these regions for each patient, which can be used for quantitative comparison.
Diffusion Tensor Imaging | Before dexmedetomidine administration
  Diffusion tensor imaging is acquired through diffusion weighted imaging (DWI)-a magnetic resonance techniques that evaluate water diffusion in terms of diffusion constants and diffusion anisotropy. From the acquired DWI, diffusion tensor imaging (DTI) allows us to model the degree of anisotropy and the structural orientation in a quantitative fashion. These DTI fractional anisotropy values will be compared pre and post-treatment.
Diffusion Tensor Imaging | Immediately following administration of dexmedetomidine
  Diffusion tensor imaging is acquired through diffusion weighted imaging (DWI)-a magnetic resonance techniques that evaluate water diffusion in terms of diffusion constants and diffusion anisotropy. From the acquired DWI, diffusion tensor imaging (DTI) allows us to model the degree of anisotropy and the structural orientation in a quantitative fashion. These DTI fractional anisotropy values will be compared pre and post-treatment.

SECONDARY OUTCOMES:
Repeatable Battery Assessment of Neuropsychological Status (RBANS) versions A-D | 1 week prior to dexmedetomidine
  RBANS assesses immediate memory, visuospatial skill, language, attention, and delayed memory. Patient performance on each subscale immediate memory, language, attention, visuospatial, and delayed memory are scored relative to validated norms for same-aged peers. A change of 8+ points in the Total Scale score, 11+ points in the Immediate Memory score, 9+ points in the Language score, 4+ points on the Attention score, 14+ points is considered significant for the Visuospatial score, and 10+ points for the Delayed Memory score are considered significant.
Quick Dementia Rating Scale (QDRS) | 1 week prior to dexmedetomidine
  The Quick Dementia Rating Scale (QDRS) is an interview-based tool administered by study officials to participants' caregivers used to obtain observations from a consistent source. The QDRS form consists of 10 categorical questions (5 cognitive, 5 functional), each with 5 detailed options depicting the level of impairment as either 0 (normal), 0.5 (mild/inconsistent impairment), 1 (mild/consistent impairment), 2 (moderate impairment), or 3 (severe impairment). Based on the conversion table outlined in Dr. James Galvin's research (2015), total QDRS scores were converted to Clinical Dementia Rating (CDR) scale levels ranging from 0 (normal aging), 0.5 (mild cognitive impairment), 1 (mild dementia), 2 (moderate dementia), and 3 (severe dementia).

CONTACTS AND LOCATIONS:
Overall Officials: Sheldon Jordan, MD, Principal Investigator — The Neurological Associates of West Los Angeles
Locations (2):
- United States (2):
  - Westwood Open MRI, Los Angeles, California
  - Neurological Associates of West Los Angeles, Santa Monica, California

IPD SHARING:
Plan to Share IPD: No
Data from this study will not be made publicly available due to ethical and privacy concerns. Anonymized data will be available upon reasonable request from any qualified investigator.

REFERENCES:
- [Background] Jagust W. Is amyloid-beta harmful to the brain? Insights from human imaging studies. Brain. 2016 Jan;139(Pt 1):23-30. doi: 10.1093/brain/awv326. Epub 2015 Nov 27. PMID 26614753
- [Background] Iliff JJ, Goldman SA, Nedergaard M. Implications of the discovery of brain lymphatic pathways. Lancet Neurol. 2015 Oct;14(10):977-9. doi: 10.1016/S1474-4422(15)00221-5. No abstract available. PMID 26376966
- [Background] Leshchyns'ka I, Liew HT, Shepherd C, Halliday GM, Stevens CH, Ke YD, Ittner LM, Sytnyk V. Abeta-dependent reduction of NCAM2-mediated synaptic adhesion contributes to synapse loss in Alzheimer's disease. Nat Commun. 2015 Nov 27;6:8836. doi: 10.1038/ncomms9836. PMID 26611261
- [Background] Thal DR, Walter J, Saido TC, Fandrich M. Neuropathology and biochemistry of Abeta and its aggregates in Alzheimer's disease. Acta Neuropathol. 2015 Feb;129(2):167-82. doi: 10.1007/s00401-014-1375-y. Epub 2014 Dec 23. PMID 25534025
- [Background] Rocha EM, De Miranda B, Sanders LH. Alpha-synuclein: Pathology, mitochondrial dysfunction and neuroinflammation in Parkinson's disease. Neurobiol Dis. 2018 Jan;109(Pt B):249-257. doi: 10.1016/j.nbd.2017.04.004. Epub 2017 Apr 8. PMID 28400134
- [Background] Lavialle M, Aumann G, Anlauf E, Prols F, Arpin M, Derouiche A. Structural plasticity of perisynaptic astrocyte processes involves ezrin and metabotropic glutamate receptors. Proc Natl Acad Sci U S A. 2011 Aug 2;108(31):12915-9. doi: 10.1073/pnas.1100957108. Epub 2011 Jul 13. PMID 21753079
- [Background] Fucke T, Suchanek D, Nawrot MP, Seamari Y, Heck DH, Aertsen A, Boucsein C. Stereotypical spatiotemporal activity patterns during slow-wave activity in the neocortex. J Neurophysiol. 2011 Dec;106(6):3035-44. doi: 10.1152/jn.00811.2010. Epub 2011 Aug 17. PMID 21849616
- [Background] Nir Y, Staba RJ, Andrillon T, Vyazovskiy VV, Cirelli C, Fried I, Tononi G. Regional slow waves and spindles in human sleep. Neuron. 2011 Apr 14;70(1):153-69. doi: 10.1016/j.neuron.2011.02.043. PMID 21482364
- [Background] de Andres I, Garzon M, Reinoso-Suarez F. Functional Anatomy of Non-REM Sleep. Front Neurol. 2011 Nov 15;2:70. doi: 10.3389/fneur.2011.00070. eCollection 2011. PMID 22110467
- [Background] Xie L, Kang H, Xu Q, Chen MJ, Liao Y, Thiyagarajan M, O'Donnell J, Christensen DJ, Nicholson C, Iliff JJ, Takano T, Deane R, Nedergaard M. Sleep drives metabolite clearance from the adult brain. Science. 2013 Oct 18;342(6156):373-7. doi: 10.1126/science.1241224. PMID 24136970
- [Background] Kress BT, Iliff JJ, Xia M, Wang M, Wei HS, Zeppenfeld D, Xie L, Kang H, Xu Q, Liew JA, Plog BA, Ding F, Deane R, Nedergaard M. Impairment of paravascular clearance pathways in the aging brain. Ann Neurol. 2014 Dec;76(6):845-61. doi: 10.1002/ana.24271. Epub 2014 Sep 26. PMID 25204284
- [Background] Mander BA, Marks SM, Vogel JW, Rao V, Lu B, Saletin JM, Ancoli-Israel S, Jagust WJ, Walker MP. beta-amyloid disrupts human NREM slow waves and related hippocampus-dependent memory consolidation. Nat Neurosci. 2015 Jul;18(7):1051-7. doi: 10.1038/nn.4035. Epub 2015 Jun 1. PMID 26030850
- [Background] Lim AS, Ellison BA, Wang JL, Yu L, Schneider JA, Buchman AS, Bennett DA, Saper CB. Sleep is related to neuron numbers in the ventrolateral preoptic/intermediate nucleus in older adults with and without Alzheimer's disease. Brain. 2014 Oct;137(Pt 10):2847-61. doi: 10.1093/brain/awu222. Epub 2014 Aug 20. PMID 25142380
- [Background] Fitzgerald PJ. Is elevated norepinephrine an etiological factor in some cases of Alzheimer's disease? Curr Alzheimer Res. 2010 Sep;7(6):506-16. doi: 10.2174/156720510792231775. PMID 20626335
- [Background] O'Donnell J, Ding F, Nedergaard M. Distinct functional states of astrocytes during sleep and wakefulness: Is norepinephrine the master regulator? Curr Sleep Med Rep. 2015 Mar;1(1):1-8. doi: 10.1007/s40675-014-0004-6. Epub 2015 Jan 29. PMID 26618103
- [Background] Plog BA, Nedergaard M. The Glymphatic System in Central Nervous System Health and Disease: Past, Present, and Future. Annu Rev Pathol. 2018 Jan 24;13:379-394. doi: 10.1146/annurev-pathol-051217-111018. PMID 29195051
- [Background] Stefanis L. alpha-Synuclein in Parkinson's disease. Cold Spring Harb Perspect Med. 2012 Feb;2(2):a009399. doi: 10.1101/cshperspect.a009399. PMID 22355802
- [Background] Shteamer JW, Dedhia RC. Sedative choice in drug-induced sleep endoscopy: A neuropharmacology-based review. Laryngoscope. 2017 Jan;127(1):273-279. doi: 10.1002/lary.26132. Epub 2016 Jul 1. PMID 27363604
- [Background] Chen K, Lu Z, Xin YC, Cai Y, Chen Y, Pan SM. Alpha-2 agonists for long-term sedation during mechanical ventilation in critically ill patients. Cochrane Database Syst Rev. 2015 Jan 6;1(1):CD010269. doi: 10.1002/14651858.CD010269.pub2. PMID 25879090
- [Background] Su X, Meng ZT, Wu XH, Cui F, Li HL, Wang DX, Zhu X, Zhu SN, Maze M, Ma D. Dexmedetomidine for prevention of delirium in elderly patients after non-cardiac surgery: a randomised, double-blind, placebo-controlled trial. Lancet. 2016 Oct 15;388(10054):1893-1902. doi: 10.1016/S0140-6736(16)30580-3. Epub 2016 Aug 16. PMID 27542303
- [Background] Seitz DP, Reimer CL, Siddiqui N. A review of epidemiological evidence for general anesthesia as a risk factor for Alzheimer's disease. Prog Neuropsychopharmacol Biol Psychiatry. 2013 Dec 2;47:122-7. doi: 10.1016/j.pnpbp.2012.06.022. Epub 2012 Jul 4. PMID 22771690
- [Background] Whittington RA, Bretteville A, Dickler MF, Planel E. Anesthesia and tau pathology. Prog Neuropsychopharmacol Biol Psychiatry. 2013 Dec 2;47:147-55. doi: 10.1016/j.pnpbp.2013.03.004. Epub 2013 Mar 25. PMID 23535147